CLINICAL TRIAL: NCT02428075
Title: Protocol for Community-based Intervention for Blood Pressure Reduction in Nepal: a Community-based Cluster Randomized Controlled Trial
Brief Title: Community-based Management of Hypertension in Nepal
Acronym: COBIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Dinesh Neupane, PhD Fellow, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hypertension-Nepal
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- FCHV visit-normotensive (Experimental)
  Interventions: Behavioral: FCHV visit
- FCHV no visit-normotensive (No Intervention)
- FCHV visit-prehypertensive (Experimental)
  Interventions: Behavioral: FCHV visit
- FCHV no visit-prehypertensive (No Intervention)
- FCHV visit-hypertensive (Experimental)
  Interventions: Behavioral: FCHV visit
- FCHV no visit-hypertensive (No Intervention)

INTERVENTIONS:
Behavioral: FCHV visit — Female Community Health Volunteer will visit selected households 3 times a year for providing health promotion messages and measure the blood pressure
  Other Names: FCHV Home Visit
  Arms: FCHV visit-hypertensive; FCHV visit-normotensive; FCHV visit-prehypertensive

SUMMARY:
Hypertension contributes to significant burden of cardiovascular diseases (CVDs) in low and middle-income countries; however responses to CVDs are inadequate particularly due to lack of conclusive evidence on population based approach to hypertension control. This is a community based cluster randomized trial involving family based health education through female community health volunteers in Nepal. People ≥25 years of age and who are listed in the voter list 2006 of Electoral Commission of Nepal who were either hypertensive, pre-hypertensive or normotensive are eligible for eligible for participation in the study. A computer generated random codes will be used to divide clusters into treatment and control arm. FCHVs will conduct family based health education and blood pressure measurements in the treatment arm vs not any interventions in control arm. Independent assessors will conduct the baseline and end line assessment of the intervention. Intention to treat analysis and per protocol analysis will be used in analysis to detect significant differences between treatment and control group participants at baseline and follow up. Student t-tests for normally distributed variables and chi-squared tests for categorical variables will be used. In the event that randomization do not control for differences between the treatment and control groups on baseline characteristics, the investigators will statistically control for those differences in subsequent analysis of program effects. The final outcome will be modeled by using multiple linear regressions analysis. The investigators hope that if the intervention outcomes shows positive effects in treatment arm, this approach can be adopted into the existing health care delivery system in Nepal. Assessing the FCHVs' ability may further contribute to developing a policy that can be scaled-up to a national level. The lessons learned from this project may also be replicated in rural areas and similar settings elsewhere in the world.

ELIGIBILITY:
Inclusion Criteria:

* People ≥25 years of age and who are listed in the voter list of 2006 and those participated in our prevalence study are eligible for inclusion in the baseline survey. - Person who give consent to participate in our intervention study,
* does not have any plan to migrate from Lekhnath Municipality for at least 1 year,
* non-pregnant women and
* personal who are not severely ill will be included as eligible participants.

Exclusion Criteria:

* No consent
* Pregnant women
* Severely Il
* Plan for migration for the study municipality within 1 year

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1638 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in mean systolic blood pressure in normotensive, pre-hypertensive and hypertensive populations | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Neupane, PhD Fellow, Principal Investigator — Center for Global Health, Aarhus University, Denmark
Locations (1):
- Lekhnath Municipality, Kāski̇̄, Gandaki, Nepal

REFERENCES:
- [Derived] Paudel S, Subedi N, McLachlan CS, Smith BJ, Kallestrup P, Neupane D. Active commuting and leisure-time physical activity among adults in western Nepal: a cross-sectional study. BMJ Open. 2021 Aug 12;11(8):e051846. doi: 10.1136/bmjopen-2021-051846. PMID 34385256
- [Derived] Neupane D, McLachlan CS, Mishra SR, Olsen MH, Perry HB, Karki A, Kallestrup P. Effectiveness of a lifestyle intervention led by female community health volunteers versus usual care in blood pressure reduction (COBIN): an open-label, cluster-randomised trial. Lancet Glob Health. 2018 Jan;6(1):e66-e73. doi: 10.1016/S2214-109X(17)30411-4. PMID 29241617
- [Derived] Neupane D, McLachlan CS, Christensen B, Karki A, Perry HB, Kallestrup P. Community-based intervention for blood pressure reduction in Nepal (COBIN trial): study protocol for a cluster-randomized controlled trial. Trials. 2016 Jun 18;17(1):292. doi: 10.1186/s13063-016-1412-3. PMID 27316539